CLINICAL TRIAL: NCT06106724
Title: Primary Precutting Versus Conventional Over-the-Wire Sphinchterotomy For Managment Of Large Common Bile Duct Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Bahaa Abdelazim, assistant lecteurer tropical medicine department sohag univerisity hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-23-09-3MD
Record Dates: First submitted 2023-10-04; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Calcular Obstructive Jaundice
MeSH Terms: interventions — Sphincterotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): sphencterotomy of papilla by conventuional methodes
  Interventions: Procedure: sphincterotomy
- group B (Active Comparator): precutting of the papilla by knife needle
  Interventions: Procedure: precutting of the papilla by knife needle

INTERVENTIONS:
Procedure: sphincterotomy — cutting the papilla and cannulation with sweeping of common bile duct by ballon and stent insertion
  Arms: group A
Procedure: precutting of the papilla by knife needle — precutting of the papilla by knife needle
  Arms: group B

SUMMARY:
During the last decades, endoscopic retrograde cholangiopancreatography (ERCP) has become the standard of care for the treatment of many pancreaticobiliary diseases [Canena et al., 2014]. However, ERCP is a challenging technique with a slow learning curve and is associated with complications, some of them lifethreatening [Chandrasekhara et al., 2017].

Post-ERCP pancreatitis (PEP) is the most common and serious complication after ERCP [Testoni et al., 2016]. A systematic survey of prospective studies including 16,885 patients reported an incidence of PEP of approximately 3.5%. Severe pancreatitis was found in 11% of the cases, and death occurred in 3% of PEP cases [Andriulli et al., 2007]. Therefore, many attempts to reduce the rate of this complication have been pursued. Selective cannulation of the common bile duct (CBD) is still considered to be a prerequisite for biliary sphincterotomy. Despite the use of various endoscopic retrograde cholangiopancreatography (ERCP) catheters and wire-guided sphincterotomes, CBD cannulation has been reported to fail in 5 % - 20 % of cases [Larkin and Huibregtse, 2001]. Precut sphincterotomy can allow access to the bile duct in such cases and is widely performed by expert endoscopists when there is a clear indication for endoscopic intervention. However, the use of precut sphincterotomy remains controversial because reported complication rates of the widely practiced needle-knife sphincterotomy (NKS) technique vary between 5 % and 20 % [Shakoor and Geenen, 1992]. Precut sphincterotomy, which includes needle-knife papillotomy (NKP), septotomy, and needle-knife fistulotomy (NKF), is often performed to facilitate access to the common bile duct of patients with difficult biliary access (DBA). Furthermore, NKF has been recommended as the preferred technique for precutting by the European Society of Gastrointestinal Endoscopy [Testoni et al., 2016] and the latest International Consensus[Liao et al., 2017]. The success of NKS also depends on the expertise of the endoscopist, and the consensus opinion is that this technique should only be performed by experienced endoscopists [Baillie,1997 ]. In contrast to NKS, incision of the papilla of Vater using an Erlangen-type precut sphincterotome has been previously reported by Binmoeller et al group to be an effective and safe auxiliary method for achieving access to the CBD after failed cannulation attempts [Binmoeller et al., 1996]. The definition of DBA varied widely [Mariani et al., 2016]. The latest guidelines for the definition of DBA differed widely from the latest guideline of The European Society of Gastrointestinal Endoscopy (defining DBA as the presence of ≥1 of the following: >5 contacts with the papilla while attempting to cannulate; >5 minutes spent attempting to cannulate following visualization of the papilla; >1 2 unintended pancreatic duct cannulation or opacification) [Testoni et al., 2016]. and the International Consensus Panel (defining DBA as the inability to achieve selective biliary cannulation by the standard ERCP technique within 10 minutes or up to 5 attempts or failure of access to the major papilla) [Liao et al., 2017 ].

ELIGIBILITY:
Inclusion Criteria:

* Patients with difficult biliary access (DBA) consenting to randomization in an interventional design randomized controlled trials (RCTs) that compare precut sphincterotomy (EPS) with persistent cannulation attempts (PCA).
* Patients who required biliary cannulation but without previous sphincterotomy.

Exclusion Criteria:

-Patients with coagulopathy or acute pancreatitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Primary Precutting Versus Conventional Over-the-Wire Sphinchterotomy For Managment Of Large Common Bile Duct Stones | 12 months
  we will assess differences between conventional sphincterotomy and primary precutting as regard which methode will be easier in cannulation, which methode wil produce more complications as acute pancreatitis, bleeding or git perforation during managment of large common bile duct stones

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Canena J, Liberato M, Coutinho AP, Marques I, Romao C, Veiga PM, Neves BC. Predictive value of cholangioscopy after endoscopic management of early postcholecystectomy bile duct strictures with an increasing number of plastic stents: a prospective study (with videos). Gastrointest Endosc. 2014 Feb;79(2):279-88. doi: 10.1016/j.gie.2013.07.022. Epub 2013 Sep 5. PMID 24012251
- [Background] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029